CLINICAL TRIAL: NCT01600820
Title: A Randomised, Double-blind, Placebo-controlled, Parallel-group Clinical Study on the Effects of a Fermented Dairy Product Enriched With Phytosterols Over Blood Cholesterol Levels of Hypercholesterolemic Adult Subjects
Brief Title: Effect of the Consumption of a Fermented Milk Enriched With Plant Sterols (Spain)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danone Spain (Industry)
Responsible Party: Sponsor
Organization: Danone Global Research & Innovation Center (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: NU146
Record Dates: First submitted 2012-05-15; First posted 2012-05-17 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Hypercholesterolemia
Keywords: Plant sterol; Hypercholesterolemia; diet; dairy; LDL-C; Mildly hypercholesterolemic subjects
MeSH Terms: conditions — Hypercholesterolemia | interventions — Phytosterols

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 = Tested product 1 (Experimental)
  Interventions: Other: 1- Low fat drinkable fermented dairy product enriched with 1.6g of plant sterol (as free equivalent) per unit
- 2 = tested product 2 (Experimental)
  Interventions: Other: 2- Low fat drinkable fermented dairy product enriched with 2.0g of plant sterol (as free equivalent) per unit
- 3 = Control product (Placebo Comparator)
  Interventions: Other: 3- Low fat drinkable fermented dairy product without plant sterols(control)

INTERVENTIONS:
Other: 1- Low fat drinkable fermented dairy product enriched with 1.6g of plant sterol (as free equivalent) per unit — 1 = Intervention 1 (1 test product/day)
  Arms: 1 = Tested product 1
Other: 2- Low fat drinkable fermented dairy product enriched with 2.0g of plant sterol (as free equivalent) per unit — 2 = Intervention 2 (1 test product/day)
  Arms: 2 = tested product 2
Other: 3- Low fat drinkable fermented dairy product without plant sterols(control) — 3 = Intervention 3 (1 control product/day)
  Arms: 3 = Control product

SUMMARY:
The purpose of this study is to investigate the cholesterol lowering effect of a drinkable low fat fermented milk enriched with plant sterol after 3 and 6 weeks in mildly hypercholesterolemic subjects treated or not by statins.

ELIGIBILITY:
Inclusion Criteria:

* male and female aged 18-75 years;
* BMI between 19 and 30 kg/m2 ,
* LDL-cholesterol higher than 130 mg/dl in individuals with a 10-year risk ≤ 20% without ischemic cardiopathy; or
* higher than 100 mg/dl in individuals with a 10-year risk > 20% or with ischemic cardiopathy (according to NCEP ATPIII guidelines),
* with or without statin monotherapy,
* willing to respect the dietary advising delivered at the screening visit,
* agreeing to a written informed consent

Exclusion Criteria:

* subject with plasma triglycerides (TG) levels > 400 mg/dL,
* with any cardiovascular event in the last 6 months,
* subject taking any drugs affecting lipid metabolism (including hypocholesterolemic treatment) other than statin in monotherapy,
* diabetic (type I and type II),
* presenting known allergy or hypersensitivity to milk proteins, soy or lactose,
* receiving systemic treatment or topical treatment likely to interfere with evaluation of the study parameters,
* with renal failure or any other metabolic disorder which could interfere with efficacy or safety assessment of the study,
* pregnant or breast feeding women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2005-02; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Sant Joan, Reus, Spain